CLINICAL TRIAL: NCT01745692
Title: A Randomised Controlled Clinical Trial of Adjunctive Mechanical Thrombectomy Compared With Intravenous Thrombolysis in Patients With Acute Ischaemic Stroke Due to an Occluded Major Intracranial Vessel.
Brief Title: Pragmatic Ischaemic Stroke Thrombectomy Evaluation
Acronym: PISTE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IDMC decision - recommended on basis of results from other relevant clinical trials, there were not safety concerns
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); University of Edinburgh (Other); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN11NE257; TSA 2011/06 (Other Grant/Funding Number: The Stroke Association)
Record Dates: First submitted 2012-11-30; First posted 2012-12-10 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Acute Ischaemic Stroke
MeSH Terms: interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous rtPA (Active Comparator): IV alteplase (rtPA) 0.9mg/kg (10% of dose as bolus followed by 90% as infusion over 1 hour, to a maximum dose of 90mg total) given within 4.5 hours of onset of stroke symptoms
  Interventions: Drug: Intravenous rtPA
- Intravenous rtPA and Mechanical Thrombectomy (Experimental): IV alteplase (rtPA) 0.9mg/kg (10% of dose as bolus followed by 90% as infusion over 1 hour, to a maximum dose of 90mg total) given within 4.5 hours of onset of stroke symptoms + additional mechanical thrombectomy procedure to commence within 90 minutes of start of IV rtPA infusion
  Interventions: Device: Mechanical thrombectomy; Drug: Intravenous rtPA

INTERVENTIONS:
Device: Mechanical thrombectomy
  Arms: Intravenous rtPA and Mechanical Thrombectomy
Drug: Intravenous rtPA — All patients receive IV alteplase
  Other Names: alteplase

SUMMARY:
Ischaemic strokes (those caused by blockage in an artery in the brain caused by a blood clot) can be treated with very early use of clot-busting (thrombolytic) drugs to attempt to restore the blood supply and limit the damage, resulting in an increased proportion of people making a recovery to independence after stroke. However, drug treatment only succeed in restoring blood flow in a minority of people with clots in the larger arteries (10-25% depending on the size of the blood vessel) and these people also have the most severe strokes and highest risk of death or dependence as a result of the stroke. Current best treatment is therefore least effective in the group with the most severe strokes. Devices that can be fed through the blood vessels to either remove or break up the blood clot in the brain vessels can open this type of large artery blockage. However, using these devices is a highly skilled procedure and it takes some time both to set up the necessary facilities (including anaesthetic, nurses and medical support) and to reach the blockage. The extra time that is required to use these devices may mean that brain tissue is already irreversibly damaged. If so, then an individual patient cannot benefit and indeed may be harmed by opening the artery. There are no completed clinical trials comparing the outcome in people treated with standard stroke treatment and those treated with devices. PISTE is a randomised, controlled trial to test whether additional mechanical thrombectomy device treatment improves functional outcome in patients with large artery occlusion who are given IV thrombolytic drug treatment as standard care.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of supratentorial acute ischaemic stroke
* Male or nonpregnant female ≥18 years of age
* Clinically significant neurological deficit and NIHSS score ≥6.
* Eligible for IV rtPA according to standard guidelines and able to be commenced on IV treatment <4.5h after symptom onset.
* Enrolment, randomisation and procedure commencement (groin puncture) possible within 90 minutes of the start of IV rtPA treatment (groin puncture maximum 5.5h after stroke onset).
* Occlusion of the main middle cerebral artery (MCA) trunk, MCA bifurcation or intracranial internal carotid artery(carotidT, M1 or single proximal M2 branch) demonstrated on CTA, MRA, or DSA.
* Interventional device delivery (guide catheter placed beyond aortic arch and angio obtained) can be achieved within 6 hours of onset of the stroke.
* Consent of patient or representative.
* Independent prior to the stroke (estimated mRS 02)
* Expected to be able to be followed up at 3 months

Exclusion Criteria:

* CT evidence of intracranial haemorrhage, or evidence of extensive established hypodensity on CT.
* Clinical history suggestive of subarachnoid haemorrhage even if CT normal.
* Known vascular access contraindications e.g. femoral bypass surgery, tight ipsilateral carotid stenosis, unsuitable proximal vascular anatomy likely to render endovascular catheterisation difficult or impossible.
* Extracranial ICA occlusion or basilar artery occlusion
* Alternative intracranial pathology potentially responsible for the new symptoms
* Medical comorbidities which would preclude safe cerebral vessel catheterisation or which are expected to limit life expectancy to <3 months (eg severe cardiac, renal or hepatic failure, significant coagulopathy, metastatic malignancy)
* Known allergy to radiological contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale | Day 90 +/-7
  The proportion with favourable functional outcome defined as mRS 0-2 at 90 (+/-7) days based on the modified Rankin scale structured interview

SECONDARY OUTCOMES:
modified Rankin Scale | Day 90+/-7
  Full neurological recovery (mRS 0-1 versus 2-6)
Mortality | Day 90 +/-7
modified Rankin Scale | Day 90 +/-7
  Change in distribution of mRS scores adjusted for baseline variables
NIH Stroke Scale (NIHSS) | 72 hours
  Early major neurological improvement of 8 or more points, or return to NIHSS total score of 0 or 1, at 72 hours (or discharge if earlier)
Angiographic patency | 22-36 hours
  Angiographic patency at 22-36 hours (Core lab assessed), using CTA or MRA
Immediate recanalisation rate | End of procedure
  Immediate (i.e. end of procedure) recanalisation rates in subjects undergoing interventional procedures (core lab assessed).
Home Time | Day 90 +/-7
  Days spent at home between stroke and day 90
Symptomatic intracranial haemorrhage | 22-26h
  Symptomatic intracranial haemorrhage rates defined as local or remote parenchymal haemorrhage type 2 (PH2 or PHr2 ICH by ECASS 2 definition) on the 22-36 h post-treatment imaging scan, combined with a neurological deterioration of 4 points or more on the NIHSS from baseline, or from the lowest NIHSS value between baseline and 24 h, or leading to death (SITS-MOST definition)
Intracranial haemorrhage | 22-36 hours
  Any intracranial haemorrhage on 22-36h CT or MRI
Significant extracranial bleeding | Up to day 90
  Extracranial bleeding, groin haematoma requiring evacuation / surgery or transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Keith W Muir, MD, FRCP, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

REFERENCES:
- [Derived] Heggie R, Wu O, White P, Ford GA, Wardlaw J, Brown MM, Clifton A, Muir KW. Mechanical thrombectomy in patients with acute ischemic stroke: A cost-effectiveness and value of implementation analysis. Int J Stroke. 2020 Oct;15(8):881-898. doi: 10.1177/1747493019879656. Epub 2019 Sep 30. PMID 31564243
- [Derived] Muir KW, Ford GA, Messow CM, Ford I, Murray A, Clifton A, Brown MM, Madigan J, Lenthall R, Robertson F, Dixit A, Cloud GC, Wardlaw J, Freeman J, White P; PISTE Investigators. Endovascular therapy for acute ischaemic stroke: the Pragmatic Ischaemic Stroke Thrombectomy Evaluation (PISTE) randomised, controlled trial. J Neurol Neurosurg Psychiatry. 2017 Jan;88(1):38-44. doi: 10.1136/jnnp-2016-314117. Epub 2016 Oct 18. PMID 27756804
- [Derived] Hurford R, Tyrrell PJ. Stroke thrombolysis: where are we and where are we going? Clin Med (Lond). 2013 Dec;13 Suppl 6:s20-3. doi: 10.7861/clinmedicine.13-6-s20. PMID 24298176